CLINICAL TRIAL: NCT04186962
Title: A Brief Intervention Involving Tetris Gameplay to Prevent Intrusive Traumatic Memories in Parents After Paediatric Intensive Care: A Feasibility Study.
Brief Title: Tetris to Reduce Intrusive Memories in Parents After PICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 262690
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2019-12

CONDITIONS: Post-traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple cognitive task (Experimental): A memory reactivation cue followed by playing the computer game "Tetris"
  Interventions: Other: Behavioral: Simple cognitive task
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Behavioral: Simple cognitive task — A memory reactivation cue followed by playing the computer game "Tetris"
  Arms: Simple cognitive task

SUMMARY:
The purpose of this study is to examine the acceptability and feasibility of a brief behavioural intervention involving Tetris gameplay to prevent intrusive traumatic memories in parents after paediatric intensive care. The present acceptability and feasibility study seeks to answer the following questions: (1) Is this intervention acceptable to parents whose children have been admitted to PICU, (2) how practical is it to deliver the intervention in this setting, (3) willingness of hospital staff to be involved in the recruitment of participants, (4) after having taken part in the intervention themselves would parents have been willing to consent to their child taking part in the intervention, and (5) discover any challenges or barriers in carrying out this study. Furthermore, this study aims to estimate recruitment, withdrawal and dropout rate, in order to act as a preliminary test of the effect of the intervention and inform sample size estimation. The findings from this study will inform the design of a randomised control trial.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child in PICU, therefore exposed to an event meeting DSM-5 criterion for a traumatic event (APA, 2013).
* The parent's child must be near the point of discharge from PICU (site 1 and 2), as identified by a clinician, or on a paediatric hospital ward within 24 hours after discharge from PICU (site 2 only).
* Sufficient ability to read and understand English to provide consent, follow game instructions and complete measures.
* Have sufficient physical mobility to play TETRIS using a computer (e.g. a handheld Nintendo DS).
* Willing and able to complete measures and be contacted one-week and month post-intervention to complete follow-up measures.

Exclusion Criteria:

* Parents will be excluded from the study if their child is due to be discharged to palliative care and/or if nursing/medical staff within the PICU feel it would be inappropriate to contact them/have them participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of flashbacks recorded by participants in a Flashback Record | Flashback Record will be returned to a researcher at one week follow-up
  The primary outcome will be the number of times a participant experiences intrusive traumatic memories related to PICU and/or the events leading to their child's admission to PICU. This will be measured using a daily pen-and-paper diary in which participants will record the occurrence of intrusive memories in everyday life for one week, starting on the day after the participant completes baseline assessment (Day 1) and completed for seven days

SECONDARY OUTCOMES:
Impact of Event Scale-Revised (IES-R) | One week and one month follow-up
  This is a self-report measure of common distressing reactions to trauma; it is comprised of three subscales, namely, intrusions, avoidance, and hyperarousal.
Pediatric Emotional Distress Scale | One week and one month follow-up
  This is a 21-item parent-report measure that assess common behaviours in young children, between 2-10 years of age, after a traumatic event.
Children's Revised Impact of Events Scale-13 Parent Version. | One week and one month follow-up
  This is a parent-report measure - Cries-13-PV.
Hospital Anxiety and Depression Scale | One week and one month follow-up
  This is a self-report questionnaire which measures anxiety and depression symptoms

OTHER OUTCOMES:
Semi-structured interviews will be conducted with participants who took part in the intervention. | Between one week and one month follow-up.
  The interview is to gain an understanding of participants views regarding being involved in the study and taking part in the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Trudie Chalder, Principal Investigator — King's College London; David McCormack, Principal Investigator — Queen's University, Belfast
Locations (2):
- United Kingdom (2):
  - Royal Belfast Hospital for Sick Children, Belfast
  - King's College London, London

IPD SHARING:
Plan to Share IPD: No